CLINICAL TRIAL: NCT05598983
Title: Non-contact Proactive Remote Monitoring to Facilitate Early Detection of Exacerbations in Chronic Obstructive Pulmonary Disease (COPD)
Brief Title: Non-contact Proactive Remote Monitoring of COPD Exacerbations
Acronym: DetectEx
Status: Recruiting | Type: Observational
Sponsor: Life Detection Technologies (Industry)
Collaborators: Royal Free Hospital NHS Foundation Trust (Other)
Responsible Party: Sponsor
Other Study IDs: DETECT EX 001
Record Dates: First submitted 2022-10-24; First posted 2022-10-31 (Actual); Last update posted 2025-03-24 (Actual); Status verified 2025-03

CONDITIONS: COPD Exacerbation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

GROUPS / COHORTS (2):
- COPD patients: Group will consist of individuals who have been diagnosed with COPD, living in their home and not recently discharged from the hospital for an exacerbation.
- Discharged COPD patients: Group will consist of individuals who have been diagnosed with COPD, living in their home, and are being discharged from the hospital for an exacerbation.

SUMMARY:
The goal of this observational study is to determine if a COPD exacerbation can be detected early in its onset. The main questions it aims to answer are:

* Can an exacerbation be detected before the person recognizes they are unwell?
* What are the biological signals which provide the best indication of decompensation?
* How does this indication of decompensation compare to a daily CAT?

Participants will be asked to place a device, DistaSense, on top of their mattress and then sleep as normal. In addition, they will be asked to complete a daily CAT.

ELIGIBILITY:
Inclusion Criteria:

1. Confirmed diagnosis of COPD
2. 1 or more exacerbation in the last year
3. Aged over 18 years
4. Willing to use monitoring devices and complete study questionnaires
5. Adequate English
6. Signed consent form

Exclusion Criteria:

1. Pregnancy
2. BMI greater than 45 kg/m2
3. Nil other, provided inclusion criteria are met.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Chronic Obstructive Pulmonary Disease (COPD) is the third leading cause of death affecting an estimated 238 million worldwide. It is a heterogeneous disease which is characterized by air flow obstruction and decline in lung function with symptoms of shortness of breathing, sputum, and cough.
Sampling Method: Non-Probability Sample
Enrollment: 75 (Estimated)
Dates: Start 2023-05-15 (Actual); Primary Completion 2026-05-15 (Estimated); Study Completion 2026-05-15 (Estimated)

PRIMARY OUTCOMES:
Track the adherence of DistaSense | 12 months
  To evaluate the adherence of patients using DistaSense, a non-contact vital sign monitor that measures heart rate and respiration rate, we will be tracking the patient dropout rate over the course of the 12 month study period.
Understand the patient acceptance of DistaSense | 12 months
  To evaluate the patient acceptance of using DistaSense, a non-contact vital sign monitor that measures heart rate and respiration rate, we will be requesting patients complete a Technology Assessment Model Fast Form (TAM-FF) every 3 months during the 12 month trial period.
Ability to detect COPD exacerbations | 3 - 12 months
  To evaluate the ability of a non-contact remote monitoring techniques to detect exacerbations of COPD.

CONTACTS AND LOCATIONS:
Overall Officials: John Hurst, Principal Investigator — University College, London
Locations (1):
- Royal Free Hospital, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No